CLINICAL TRIAL: NCT01192464
Title: Phase I Study of the Administration of EBV CTLs Expressing CD30 Chimeric Receptors for Relapsed CD30+ Hodgkin's Lymphoma and CD30+ Non-Hodgkin's Lymphoma (CAR CD 30)
Brief Title: EBV CTLs Expressing CD30 Chimeric Receptors For CD 30+ Lymphoma
Acronym: CARCD30
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-26617 CAR CD 30
Record Dates: First submitted 2010-08-16; First posted 2010-09-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- autologous CAR.CD30 EBV specific-CTLs (Experimental): Group One Dose (CTLs CAR.CD30) at Day 0: 2x10^7 cells/m2
  Group Two Dose (CTLs CAR.CD30) at Day 0: 5x10^7 cells/m2
  Group Three Dose (CTLs CAR.CD30) at Day 0: 1x10^8 cells/m2
  Interventions: Drug: autologous CAR.CD30 EBV specific-CTLs

INTERVENTIONS:
Drug: autologous CAR.CD30 EBV specific-CTLs — Three dose levels will be evaluated. Using the modified continual reassessment method, cohorts of size two will be enrolled at each dose level. Each patient will receive one injection.
  Other Names: CD30 EBV CTL

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins the protect the body from diseases caused by germs or toxic substances. They work by binding those germs or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with germs. Both antibodies and T cells have been used to treat patients with cancers: they both have been shown promise, but have not been strong enough to cure most patients. This study combines the two methods.

We have found from previous research that we can put a new gene into T cells that will make them recognize cancer cells and kill them. We now want to see if we can attach a new gene to T cells that will help them do a better job at recognizing and killing lymphoma cells.

The new gene we will put in T cells makes an antibody called anti-CD30. The antibody alone has not been strong enough to cure most patients. For this study, the anti-CD30 antibody has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These chimeric receptor-T cells seem to kill some of the tumor, but they don't last very long and so their chances of fighting the cancer are unknown.

We have found that T cells that are also trained to recognize the EBV virus (that causes infectious mononucleosis) can stay in the blood stream for many years. These are called EBV specific Cytotoxic T Lymphocytes.

By joining the anti-CD30 antibody to the EBV CTLs, we believe that we will also be able to make a cell that can last a long time in the body and recognize and kill lymphoma cells. We call the final cells CD30 chimeric receptor EBV CTLs. T

We hope that these new cells may be able to work longer and target and kill lymphoma cells. However, we do not know that yet.

DETAILED DESCRIPTION:
The EBV CTLs will be made for specific patients. First blood will be collected from the patient and then the the CD30 chimeric-EBV CTLs will be created in the lab. The cells will then be grown and frozen for the patient.

To get the CD30 antibody to attach to the surface of the T cell, the lab will insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. Because the patient will have received cells with a new gene in them they will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When the patient is enrolled on this study, they will be assigned to one of the following dose levels of CD30 chimeric receptor-EBV CTLs.

* 2×10^7 cells/m2
* 5x10^7 cells/m2
* 1×10^8 cells/m2

The dose level of cells that they will receive will not be based on a medical determination of what is best for them, instead the dose is based on the order in which the patient enrolls on the study relative to other participants. Subjects enrolled earlier in the study will receive a lower dose of cells than those enrolled later in the study. The risks of harm and discomfort from the study treatment may bear some relationship to the dose level. The potential for direct benefit, if any, may also vary with the dose level. To enroll on this study they will need to have recovered from toxic effects of previous chemotherapy for at least one week and not be receiving any other investigational agents. Patients cannot have received any tumor vaccines within the previous six weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

PROCUREMENT Inclusion Criteria:

* Referred patients will initially be consented for procurement of blood for generation of the transduced CTL Line. Eligibility criteria at this stage include:
* Diagnosis of recurrent HL or NHL, or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory HL or NHL with a treatment plan that will include high dose therapy and stem cell transplantation
* CD30 positive tumor (can be pending at this time)
* EBV seropositivity (can be pending at this time)
* Hgb > 8.0
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

TREAMENT Inclusion Criteria: Patients must meet the following eligibility criteria to be included for treatment:

* Diagnosis - CD30+ HL or CD30+ NHL
* During the dose escalation phase: only adult patients (age 18 and older) with active disease failing standard therapy
* After dose escalation: any patient (children or adults) with relapsed CD30+ HL or CD30+ NHL or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory CD30+ HL or CD30+ NHL with a treatment plan that will include high dose therapy and autologous stem cell transplantation.
* CD30 positive tumor
* EBV seropositivity.
* Recovered from acute toxic effects of all prior chemotherapy at least one week and 30 days from prior chemotherapy before entering this study.
* Bilirubin 1.5 times or less than upper limit of normal.
* AST 3 times or less than upper limit of normal.
* Serum creatinine 1.5 times or less than upper limit of normal.
* Pulse oximetry of > 90% on room air
* Karnofsky or Lansky score of > 60%.
* Available autologous transduced EBV-specific cytotoxic T lymphocytes with 15% or more expression of CD30CAR determined by flow-cytometry.
* Adequate pulmonary function with FEV1, FVC and DLCO 50% or greater of expected corrected for hemoglobin. Exceptions may be allowed for patients with pulmonary involvement after discussing with PI.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

EXCLUSION CRITERIA:

PROCUREMENT Exclusion Criteria:

* Active infection with HIV, HTLV, HBV, HCV (can be pending at this time).
* Received rituximab within 4 months of blood collection for LCL initiation (unless circulating CD19+ B are =/>2%)

TREATMENT Exclusion Criteria:

* Currently receiving any investigational agents or received any tumor vaccines within the previous six weeks.
* Received anti-CD30 antibody-based therapy within the previous 6 weeks.
* History of hypersensitivity reactions to murine protein-containing products.
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Current use of systemic corticosteroids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-05-10 (Actual); Primary Completion 2012-05-29 (Actual); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of escalating doses of autologous EBV-specific cytotoxic T-lymphocytes (CTLs), | 6 weeks
  To evaluate the safety of escalating doses of autologous EBV-specific cytotoxic T-lymphocytes (CTLs), genetically modified to express an artificial T-cell receptor (CAR) targeting the CD30 molecule (CAR.CD30), in patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL)

SECONDARY OUTCOMES:
To measure the survival of CAR.CD30 transduced EBV-CTLs in vivo. | 15 years
  To measure the survival of CAR.CD30 transduced EBV-CTLs in vivo.
To measure the anti-tumor effects of CAR.CD30 transduced CTLs | 8 weeks
  To measure the anti-tumor effects of CAR.CD30 transduced CTLs in patients with patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL)

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine/Center for Cell and Gene Therapy
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT01192464/ICF_000.pdf